CLINICAL TRIAL: NCT00947427
Title: Effects of Canakinumab On The Progression of Type 1 Diabetes In New Onset Subjects
Brief Title: Canakinumab Study in Individuals With Newly Diagnosed Type 1 Diabetes
Acronym: TN14
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TN14 Cana; UC4DK097835 (NIH)
Record Dates: First submitted 2009-07-24; First posted 2009-07-28 (Estimated); Results first posted 2016-10-18 (Estimated); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Type 1 Diabetes; Preservation of Insulin Secretion; Newly Diagnosed Type 1 Diabetes; Canakinumab in Type 1 Diabetes
Keywords: type 1 diabetes; newly diagnosed T1D; T1D; canakinumab; anti IL-1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — canakinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo solution given by subcutaneous injection on monthly basis for 12 months
  Interventions: Drug: Placebo
- Canakinumab (Experimental): Subcutaneous injection of canakinumab at dose of 2.0 mg/kg given monthly of 12 months
  Interventions: Drug: canakinumab (anti IL-1beta)

INTERVENTIONS:
Drug: canakinumab (anti IL-1beta) — canakinumab subcutaneous injections given at 2.0mg/kg dose on monthly basis for 12 months
  Other Names: canakinumab; anti IL-1beta
  Arms: Canakinumab
Drug: Placebo — Placebo subcutaneous injections
  Arms: Placebo

SUMMARY:
Canakinumab is a fully human anti-interleukin-1β (anti-IL-1β) monoclonal antibody (IgG-1 class). Canakinumab is designed to bind to human IL-1β and to functionally neutralize the bioactivity of this pro-inflammatory cytokine.

The study is a two-arm, multicenter, randomized, double-masked, placebo-controlled clinical trial. 66 subjects will be randomly assigned to receive either monthly subcutaneous injections of 2.0 mg/kg Canakinumab, or placebo for 12 months. All groups will receive standard intensive diabetes treatment with insulin and dietary management.

Participants randomly assigned to Canakinumab treatment or placebo will receive a total of 12 injections over one year.

All subjects will be followed for 1 year of treatment plus 1- 3 years of additional follow-up until study end. Enrollment is expected to occur over two years.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 6-45 years
* Be within 3-months (100 days) of diagnosis of type 1 diabetes
* Must have at least one diabetes-related autoantibody present
* Must have stimulated C-peptide levels >0.2 pmol/ml measured during a mixed meal tolerance test (MMTT) conducted at least 21 days from diagnosis and within 37 days of randomization
* If participant is female with reproductive potential, she must be willing to avoid pregnancy and have a negative pregnancy test during the 12 months of treatment and for an additional 3 months after completing treatment
* Be at least one month from time of last live immunization received
* Willing to forgo live vaccinations for 24 months
* Must be willing to comply with intensive diabetes management
* Must weigh at least 20 kg (44 lbs) at study entry

Exclusion Criteria:

* Are immunodeficient or have clinically significant chronic lymphopenia (low white blood cell count)
* Have an active infection
* Have a positive PPD test result
* Be currently pregnant or lactating, or anticipate getting pregnant
* Ongoing use of medications known to influence glucose tolerance
* Require use of other immunosuppressive agents
* Have serologic evidence of current or past HIV, Hepatitis B, or Hepatitis C infection
* Have any complicating medical issues or abnormal clinical laboratory blood counts or results that interfere with study conduct; history of malignancies
* Be currently participating in another type 1 diabetes treatment study

Ages: 6 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 71 (Actual)
Dates: Start 2010-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (11):
  - University of California-San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Yale Medical School, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Indiana University-Riley Hospital for Children, Indianapolis, Indiana
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas-Southwestern Medical School, Dallas, Texas
  - Benaroya Research Institute, Seattle, Washington
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data are available at the NIDDK Central Repository:https://repository.niddk.nih.gov/studies/tn14-anti-il-1-beta/?query=TN14
URL: https://repository.niddk.nih.gov/studies/tn14-anti-il-1-beta/?query=TN14

REFERENCES:
- [Result] Moran A, Bundy B, Becker DJ, DiMeglio LA, Gitelman SE, Goland R, Greenbaum CJ, Herold KC, Marks JB, Raskin P, Sanda S, Schatz D, Wherrett DK, Wilson DM, Krischer JP, Skyler JS; Type 1 Diabetes TrialNet Canakinumab Study Group; Pickersgill L, de Koning E, Ziegler AG, Boehm B, Badenhoop K, Schloot N, Bak JF, Pozzilli P, Mauricio D, Donath MY, Castano L, Wagner A, Lervang HH, Perrild H, Mandrup-Poulsen T; AIDA Study Group. Interleukin-1 antagonism in type 1 diabetes of recent onset: two multicentre, randomised, double-blind, placebo-controlled trials. Lancet. 2013 Jun 1;381(9881):1905-15. doi: 10.1016/S0140-6736(13)60023-9. Epub 2013 Apr 5. PMID 23562090

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Injection: Placebo solution (2.0/kg dose) given subcutaneously on monthly basis for 12 months
Period: Overall Study
Arm/Group | Placebo Injection | Canakinumab (Anti IL-1beta)
Started | 22 | 49 (2 participants discontinued prior to any study drug administration)
Completed | 21 | 45
Not Completed | 1 | 4
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Injection | Canakinumab (Anti IL-1beta) | Total
Number analyzed (Participants) | 22 | 49 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.4 (6.4) | 11.6 (4.0) | 11.8 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 25 | 33
  Male | 14 | 24 | 38

OUTCOME MEASURES:

1. Primary Outcome: C-peptide Response to Mixed Meal Glucose Tolerance Test (MMTT) at One Year for Subjects Given Canakinumab Compared to Placebo
Description: The primary outcome is the area under the stimulated C-peptide curve (AUC) based on data collected at time 0 to 2 hours of a 4-hour mixed meal glucose tolerance test (MMTT) conducted at the primary endpoint visit. The timed measurements are done at: 0, 15, 30 60, 90, and 120 minutes. The calculation for the concentration of c-peptide is a weighted average of the 6 timed measurements of c-peptide in nano-moles/Liter. We try to distinguish this calculation from the AUC by referring to it as the "AUC mean" and may be expressed algebraically as the AUC/(120 min.); thus, the units are the same as the y-axis.
Time Frame: 12 months
Measure: Geometric Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Placebo Injection | Canakinumab (Anti IL-1beta)
Number analyzed (Participants) | 21 | 45
nmol/L | 0.40 [0.30 to 0.49] | 0.41 [0.34 to 0.47]
Statistical Analysis 1: Comparison: Placebo Injection vs Canakinumab (Anti IL-1beta); Test type: Superiority or Other; p = 0.86, ANCOVA

ADVERSE EVENTS:
Arm/Group | Placebo Injection | Canakinumab (Anti IL-1beta)
Serious Adverse Events (participants affected / at risk) | 1/22 | 1/49
Other Adverse Events (participants affected / at risk) | 15/22 | 30/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Injection (N=22) | Canakinumab (Anti IL-1beta) (N=49)
Endocrine - Other (Endocrine disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Injection (N=22) | Canakinumab (Anti IL-1beta) (N=49)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 3 (7) | 8 (12)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (6)
Vomiting (Gastrointestinal disorders) | 3 (4) | 3 (3)
Infection - Other (Infections and infestations) | 6 (10) | 7 (9)
Infection with unknown ANC- Middle ear (otitis media) (Infections and infestations) | 1 (2) | 3 (4)
Infection with unknown ANC- Pharynx (Infections and infestations) | 2 (2) | 5 (5)
Infection with unknown ANC- Sinus (Infections and infestations) | 1 (1) | 4 (5)
Infection with unknown ANC- Skin (cellulitis) (Infections and infestations) | 3 (3) | 3 (4)
Infection with unknown ANC- Upper airway (Infections and infestations) | 3 (3) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Pain - Other (General disorders) | 2 (3) | 4 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No